CLINICAL TRIAL: NCT02079233
Title: Phase 1 Multiple Dose Trial to Assess the Safety, Tolerability and Efficacy of Four Different Dosing Regimens of Cross-Linked Polyelectrolyte (CLP) in Healthy Volunteers
Brief Title: Evaluation of Four Different Dosing Regimens of Cross-Linked Polyelectrolyte (CLP) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorbent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTST-16
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Basic Science; Safety; Tolerability; Efficacy of CLP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CLP 15 g QD (Experimental): Cross-Linked Polyelectrolyte (CLP) study medication delivered immediately before bedtime
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)
- CLP 7.5 g BID (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered b.i.d. one hour before breakfast and dinner
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)
- CLP 5 g TID (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered t.i.d. one hour before breakfast, lunch and dinner
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)
- CLP 3.75 g QID (Experimental): Cross-Linked Polyelectrolyte (CLP) Study medication delivered q.i.d on hour before breakfast, lunch, dinner and immediately before bedtime
  Interventions: Drug: Cross-Linked Polyelectrolyte (CLP)

INTERVENTIONS:
Drug: Cross-Linked Polyelectrolyte (CLP) — CLP was administered orally, in capsules, for 7 consecutive days.

SUMMARY:
This is a study to determine the effect of four different dosing regimens of CLP in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer is ≥ 18 years of age with BMI of 18-32
* Females could not be pregnant or breast feeding and had to be using birth control
* Must have regular bowel habits, typically producing at least 1 daily bowel movement

Exclusion Criteria:

* Screening 12-lead ECG demonstrating QTc interval >430 msec for males and >450 msec for females, or any cardiac rhythm disorder considered by the Investigator to be clinically relevant
* History or presence of gastrointestinal conditions
* Positive drug screen for substances of abuse
* Positive results for HIV, hepatitis B, or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in fecal sodium content | Baseline (Days 3-6) vs. Treatment (Days 10-13)
  The primary endpoint was sodium removal from the stool compared between the Baseline period and the Treatment Period.

CONTACTS AND LOCATIONS:
Overall Officials: Shanthini A. Daniel, MD, Principal Investigator — Jasper Clinic, Inc.